CLINICAL TRIAL: NCT02620007
Title: Multicenter Double Blind Randomized Clinical Trial Assessing the Benefit of Adherent Invasive E. Coli Eradication in Adult Ileal and Ileo-colonic Crohn Disease
Brief Title: Evaluation of Adherent Invasive E. Coli Eradication in Adult Crohn Disease
Acronym: TEOREM
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P140503
Record Dates: First submitted 2015-11-30; First posted 2015-12-02 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2019-02

CONDITIONS: Crohn Disease; Adherent-invasive E. Coli
Keywords: Adult; AIEC
MeSH Terms: conditions — Crohn Disease | interventions — Ciprofloxacin; Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): oral Ciprofloxacin 500 mg bid and oral Rifaximin 800 mg bid for 12 weeks
  Interventions: Drug: Ciprofloxacin; Drug: Rifaximin
- Control arm (Placebo Comparator): a placebo of Ciprofloxacin bid and a placebo of Rifaximin bid for 12 weeks
  Interventions: Drug: Ciprofloxacin Placebo; Drug: Rifaximin Placebo

INTERVENTIONS:
Drug: Ciprofloxacin — oral Ciprofloxacin 500 mg bis in die (bid) for 12 weeks
  Arms: Experimental arm
Drug: Rifaximin — oral Rifaximin 800 mg bid for 12 weeks
  Arms: Experimental arm
Drug: Ciprofloxacin Placebo — a placebo of Ciprofloxacin bid for 12 weeks
  Arms: Control arm
Drug: Rifaximin Placebo — a placebo of Rifaximin bid for 12 weeks
  Arms: Control arm

SUMMARY:
The primary objective of this trial is to assess whether a 12-week treatment with Ciprofloxacin and Rifaximin is superior to placebo to obtain endoscopic remission in adherent-invasive E. coli (AIEC)-colonized patients with ileal Crohn disease (CD), with or without involvement of the caecum or the right colon.

ELIGIBILITY:
Inclusion Criteria:

* CD of the ileum, with or without involvement of the caecum or the right colon
* Colonoscopy showing active lesions defined by a CDEISm score >6
* Informed consent to participate in this study
* Prescription of steroid treatments : Budesonide, Prednisone (or Prednisolone) independently from entry in study
* Patients who respond to budesonide (initial dose 9 mg/d) or prednisone or prednisolone (initial dose 40 mg/d), defined as a 70 points decrease in CDAI between the pre-inclusion and the inclusion visit,
* Patients colonized with AIEC on initial ileal biopsies.

Exclusion Criteria:

* Ileal stenosis that cannot be crossed by the endoscope,
* Infliximab treatment received less than 8 weeks before inclusion in this study,
* Adalimumab treatment received less than 4 weeks before inclusion in this study,
* Vedolizumab treatment received less than 8 weeks before inclusion in the study,
* Hypersensitivity to Ciprofloxacin, to other quinolones, or to any of the excipients (cellulose microcrystalline, crospovidone, maize starch, magnesium stearate, silica colloidal anhydrous,, hypromellose titanium dioxide E171, macrogol 4000,),
* Tizanidine, Probenecid, Theophylline, Xanthine derivatives, Phenytoin, oral anticoagulants, and Ropinirole treatment,
* Hypersensitivity to Rifaximin, or to any excipients (sodium starch glycolate type A, glycerol distearate, colloidal anhydrous silica, talc, microcrystalline cellulose, hypromellose, titanium dioxide, disodium edentate, propylene glycol, red iron oxide E172),
* Previous extensive ileal surgery (≥ 1 meter as measured on the pathology and/or surgical report),
* Short bowel syndrome,
* Need for an intestinal resection for fistula, abscess or intestinal obstruction,
* Renal failure (creatinine clearance<30 mL/min/1.73m2),
* Liver failure (V factor<50%),
* Past history of epilepsy,
* No health insurance,
* Pregnant or lactating women,
* Refusal to have a double effective contraception,
* Patients already included in a biomedical research other than an observational study (e.g: registry, cohort).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12; Primary Completion 2021-08 (Actual); Study Completion 2022-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with Endoscopic Endoscopic Index of Severity (CDEISm)< 6 and a decrease in CDEISm ≥ 3 | week 12
  (assessed within each site quotation), defined by the modified Crohn's Disease Endoscopic Index of Severity (CDEISm)< 6 and a decrease in CDEISm ≥ 3, as compared to baseline values.

SECONDARY OUTCOMES:
Mean variation of CDEISm | week 12
  assessed by centralized, anonymous and blinded reading of ileocolonoscopies
Complete endoscopic remission | week 12
  assessed by centralized, anonymous and blinded reading of ileocolonoscopies, and defined by a CDEISm <3
No ulceration | week 12
Clinical remission | 12 and 48 weeks
  defined by Crohn's disease activity index (CDAI)<150 without steroids, anti-Tumor Necrosis Factor (TNF), and surgery
Microbiota composition | weeks 12 and 48
lpf positive AIEC bacteria in the stools | weeks 12 and 48
  Detection (by PCR)
Biological remission | weeks 4, 8, 12, 24, 36 and 48
  defined by haemoglobin level ≥13g/dL and C-Reactive Protein (CRP) serum level ≤5 mg/L and fecal calprotectin <300 mg/L
Side effects | week 12
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Barnich, MD PhD, Study Chair — Intestinal bacterial pathogenesis laboratory
Locations (2):
- France (2):
  - Kremlin-Bicetre hospital, Le Kremlin-Bicêtre
  - Gastroenterology department, Le Kremlin-Bicêtre